CLINICAL TRIAL: NCT06348836
Title: The Effects of Open Chain Versus Closed Chain Strengthening on Dynamic Valgus During a Step Down Test
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alvernia University (Other)
Responsible Party: Principal Investigator, James O'Donohue, Associate Professor of Physical Therapy, Alvernia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2123624-1/2
Record Dates: First submitted 2024-03-30; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Dynamic Knee Valgus
Keywords: knee valgus; hip weakness
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either a closed-chain (weightbearing) exercise group or an open-chain (non-weightbearing) exercise group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed-Chain exercise (Active Comparator): 4 exercises: 1)Single leg bridge, 2)side plank (with testing side down), 3) single leg squat, 4) banded squat Exercises to be performed with 3 sets of 10 repetitions each. Frequency will be 2 times per week for 6 weeks.
  Interventions: Other: Exercise
- Open-Chain exercise (Active Comparator): 4 exercises: 1) Side plank (with testing side up), 2) clamshells, 3) front plank with hip extension, 4)wall slide Exercises to be performed with 3 sets of 10 repetitions each. Frequency will be 2 times per week for 6 weeks.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Description of exercises are noted in the arms/groups descriptions
  Other Names: Closed-chain exercise; Open-chain exercise

SUMMARY:
The goal of this clinical trial is to compare the effects of different exercises programs in individuals with abnormal knee motion. The main question it aims to answer are:

* In individuals with abnormal knee motion and without knee pain, does a weight-bearing exercise program reduce abnormal knee motion during a step-down test better than a non weight-bearing exercise program? Participants will
* Perform a stepdown test while undergoing motion analysis and electromyograph (EMG) recording.
* Participants will then be placed either into a weight-bearing or non weight-bearing exercise group. Exercises will be performed 3 times per week for 6 weeks.
* Further motion analysis and EMG data will be collected to test for differences. Researchers will compare individual results before and after exercise, and between-group results before and after exercise to see if one exercise program helps improved abnormal knee motion more than the other.

DETAILED DESCRIPTION:
The goals of this trial is to compare the effects of a closed kinetic chain exercise program to an open kinetic chain exercise program in individuals without knee pain who also have dynamic knee valgus during a step-down test.

Individuals will be screened for participation via visual observation. Those with an observable medial collapse of the knee joint will then receive motion capture testing of the step down test (three trials) with electromyography recording of the gluteus medius, quadriceps and hamstring muscle groups. Baseline maximum voluntary contraction of these muscles will be done with EMG analysis and force gauge measurements.

After initial data collection participants will be randomized into either a closed kinetic chain exercise group or open kinetic chain exercise group. (described in the Arms section) Participants will exercise 2-3 times per week for 6 weeks. After the exercise program is completed, participants will then be seen back for final data collection which will match the initial collection process.

ELIGIBILITY:
Inclusion Criteria:

* Dynamic knee valgus with observed step down test

Exclusion Criteria:

* Presently experiencing lower extremity pain
* Lower extremity surgery within the past 1 year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Electromyographic activity of gluteus medius muscle during step-down test | 6 weeks
  Muscle activity of gluteus medius during max contraction and during step-down test
Electromyographic activity of quadriceps muscle during step-down test | 6 weeks
  Muscle activity of quadriceps muscle during max contraction and during step-down test
Electromyographic activity of hamstring muscles during step-down test | 6 weeks
  Muscle activity of hamstring muscles during max contraction and during step-down test

SECONDARY OUTCOMES:
Amount of dynamic knee valgus during step-down test measured with motion analysis | 6 weeks
  Motion analysis of frontal plane knee motion during step-down test

CONTACTS AND LOCATIONS:
Overall Officials: James M O'Donohue, DPT, Principal Investigator — Alvernia University
Locations (1):
- Alvernia University, Reading, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data at this time

REFERENCES:
- [Background] Devereaux MD, Lachmann SM. Patello-femoral arthralgia in athletes attending a Sports Injury Clinic. Br J Sports Med. 1984 Mar;18(1):18-21. doi: 10.1136/bjsm.18.1.18. PMID 6722419
- [Background] Bunt CW, Jonas CE, Chang JG. Knee Pain in Adults and Adolescents: The Initial Evaluation. Am Fam Physician. 2018 Nov 1;98(9):576-585. PMID 30325638
- [Background] Fukuda TY, Rossetto FM, Magalhaes E, Bryk FF, Lucareli PR, de Almeida Aparecida Carvalho N. Short-term effects of hip abductors and lateral rotators strengthening in females with patellofemoral pain syndrome: a randomized controlled clinical trial. J Orthop Sports Phys Ther. 2010 Nov;40(11):736-42. doi: 10.2519/jospt.2010.3246. PMID 21041965
- [Background] Bolgla LA, Boling MC, Mace KL, DiStefano MJ, Fithian DC, Powers CM. National Athletic Trainers' Association Position Statement: Management of Individuals With Patellofemoral Pain. J Athl Train. 2018 Sep;53(9):820-836. doi: 10.4085/1062-6050-231-15. PMID 30372640
- [Background] Dutton RA, Khadavi MJ, Fredericson M. Patellofemoral Pain. Phys Med Rehabil Clin N Am. 2016 Feb;27(1):31-52. doi: 10.1016/j.pmr.2015.08.002. PMID 26616176
- [Background] Hollman JH, Ginos BE, Kozuchowski J, Vaughn AS, Krause DA, Youdas JW. Relationships between knee valgus, hip-muscle strength, and hip-muscle recruitment during a single-limb step-down. J Sport Rehabil. 2009 Feb;18(1):104-17. doi: 10.1123/jsr.18.1.104. PMID 19321910
- [Background] Stickler L, Finley M, Gulgin H. Relationship between hip and core strength and frontal plane alignment during a single leg squat. Phys Ther Sport. 2015 Feb;16(1):66-71. doi: 10.1016/j.ptsp.2014.05.002. Epub 2014 Jun 3. PMID 25070759
- [Background] Scholtes SA, Salsich GB. A DYNAMIC VALGUS INDEX THAT COMBINES HIP AND KNEE ANGLES: ASSESSMENT OF UTILITY IN FEMALES WITH PATELLOFEMORAL PAIN. Int J Sports Phys Ther. 2017 Jun;12(3):333-340. PMID 28593087
- [Background] Chowdhury RH, Reaz MB, Ali MA, Bakar AA, Chellappan K, Chang TG. Surface electromyography signal processing and classification techniques. Sensors (Basel). 2013 Sep 17;13(9):12431-66. doi: 10.3390/s130912431. PMID 24048337
- [Background] Harris-Hayes M, Steger-May K, Koh C, Royer NK, Graci V, Salsich GB. Classification of lower extremity movement patterns based on visual assessment: reliability and correlation with 2-dimensional video analysis. J Athl Train. 2014 May-Jun;49(3):304-10. doi: 10.4085/1062-6050-49.2.21. PMID 24955621
- [Background] Simon M, Parizek C, Earl-Boehm JE, Bazett-Jones DM. Quantitative and qualitative assessment of frontal plane knee motion in males and females: A reliability and validity study. Knee. 2018 Dec;25(6):1057-1064. doi: 10.1016/j.knee.2018.09.008. Epub 2018 Nov 8. PMID 30414788
- [Background] Kunene SH, Taukobong NP, Ramklass S. Rehabilitation approaches to anterior knee pain among runners: A scoping review. S Afr J Physiother. 2020 Jan 27;76(1):1342. doi: 10.4102/sajp.v76i1.1342. eCollection 2020. PMID 32161824
- [Background] Ismail MM, Gamaleldein MH, Hassa KA. Closed kinetic chain exercises with or without additional hip strengthening exercises in management of patellofemoral pain syndrome: a randomized controlled trial. Eur J Phys Rehabil Med. 2013 Oct;49(5):687-98. Epub 2013 Jul 2. PMID 23820880
- [Background] Moore D, Semciw AI, Pizzari T. A SYSTEMATIC REVIEW AND META-ANALYSIS OF COMMON THERAPEUTIC EXERCISES THAT GENERATE HIGHEST MUSCLE ACTIVITY IN THE GLUTEUS MEDIUS AND GLUTEUS MINIMUS SEGMENTS. Int J Sports Phys Ther. 2020 Dec;15(6):856-881. doi: 10.26603/ijspt20200856. PMID 33344003
- [Background] Boren K, Conrey C, Le Coguic J, Paprocki L, Voight M, Robinson TK. Electromyographic analysis of gluteus medius and gluteus maximus during rehabilitation exercises. Int J Sports Phys Ther. 2011 Sep;6(3):206-23. PMID 22034614
- [Background] Willy RW, Davis IS. The effect of a hip-strengthening program on mechanics during running and during a single-leg squat. J Orthop Sports Phys Ther. 2011 Sep;41(9):625-32. doi: 10.2519/jospt.2011.3470. Epub 2011 Jul 12. PMID 21765220